CLINICAL TRIAL: NCT00800618
Title: A Double Blind (3rd Party Open), Randomised, Placebo Controlled, Dose Escalating, Parallel Group Study To Investigate The Safety, Toleration, Pharmacology And Pharmacokinetics, Of Multiple Doses Of PF-02413873 In Healthy Female Subjects.
Brief Title: A Study To Investigate How The Body Handles Multiple Doses Of PF-0243873 And To Investigate The Effect Of PF-02413873 On Sex Hormone Levels In Healthy Young Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B0461002
Record Dates: First submitted 2008-12-01; First posted 2008-12-02 (Estimated); Last update posted 2010-02-10 (Estimated); Status verified 2010-02

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — 4-(3-cyclopropyl-1-(methylsulfonylmethyl)-5-methyl-1H-pyrazol-4-yl)oxy-2,6-dimethylbenzonitrile

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-02413873 (Experimental): PF-2413873 active treatment
  Interventions: Drug: PF-02413873 100 mg QD; Drug: PF-02413873 1500 mg QD; Drug: PF-02413873 20 mg QD; Drug: PF-02413873 500 mg QD
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: PF-02413873 Placebo

INTERVENTIONS:
Drug: PF-02413873 100 mg QD — 100 mg of PF-02413873 oral suspension once daily for 14 days
  Arms: PF-02413873
Drug: PF-02413873 1500 mg QD — 1500 mg of PF-02413873 oral suspension once daily for 14 days
  Arms: PF-02413873
Drug: PF-02413873 20 mg QD — 20 mg of PF-02413873 oral suspension once daily for 14 days
  Arms: PF-02413873
Drug: PF-02413873 500 mg QD — 500 mg of PF-02413873 oral suspension once daily for 14 days
  Arms: PF-02413873
Drug: PF-02413873 Placebo — PF-0241383 Placebo once daily for 14 days
  Arms: Placebo

SUMMARY:
The study will investigate how well multiple doses of PF-02413873 are tolerated by healthy young women, how the body handles multiple doses of PF-02413873 and which effect PF-02413873 has on sex hormones in healthy young women

ELIGIBILITY:
Inclusion Criteria:

* Healthy women of childbearing potential with a regular menstrual cycle

Exclusion Criteria:

* Evidence or history of any major disease
* Pregnant or nursing women
* Requirement for chronic medication

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2008-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Adverse events, vital signs measurements, 12-lead ECGs, physical examination findings, blood safety tests. | 1 month
PF-02413873 pharmacokinetics | 1 month
Endometrial thickness, Ovarian follicular estradiol secretion, Pre-ovulatory LH surge, Corpus Luteum progesterone secretion. | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (2):
  - Pfizer Investigational Site, New Haven, Connecticut
  - Pfizer Investigational Site, Overland Park, Kansas
- Pfizer Investigational Site, Brussels, Belgium